CLINICAL TRIAL: NCT03188250
Title: Increasing Pregnancy Health Services Uptake Through Integrated Peer Support Groups in Kenya: A Prospective Cohort Study
Brief Title: Chama Cha MamaToto: a Pilot Study of Peer Support Groups in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moi University (Other)
Collaborators: Grand Challenges Canada (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Astrid Christoffersen-Deb, Visiting Lecturer, Moi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMoi3
Record Dates: First submitted 2017-05-31; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy Related; Group, Peer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chama cha MamaToto (Experimental): Pregnant women in communities where chama cha mamatoto is taking place will be invited to join and participate in bi-weekly group meetings for a year
  Interventions: Behavioral: Chama cha Mamtoto
- Referent (No Intervention): Pregnant women attending at least one prenatal visit in communities where chama cha mamatoto was implemented three months later served as the comparison

INTERVENTIONS:
Behavioral: Chama cha Mamtoto — Chama cha Mamatoto is a community-based model of peer support group in pregnancy and infancy that combines health education, relationship building and a savings and loans program, led by community health workers
  Arms: Chama cha MamaToto

SUMMARY:
Preventing maternal and newborn deaths remain high on the global agenda. To address this, the Academic Model Providing Access to Healthcare (AMPATH), in partnership with the Government of Kenya, launched Chama cha MamaToto, a community-led peer-support model that groups women together in pregnancy and infancy. Central to the chama approach is the integration of health, social and financial literacy education with a savings/loans program.

DETAILED DESCRIPTION:
To evaluate the feasibility of chamas, we analysed group attendance rates, GISE participation, membership retention, and continuation of the groups beyond the one year. To evaluate the effect of chamas, the investigators compared data from a prospective cohort of women in chamas with a group of controls who did not belong to a chama, matched for age, parity, and location of prenatal care. To evaluate the acceptability of chamas, FGDs were carried out with chama and non-chama participants, health providers and community health workers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in communities where chamas were taking place
* Any woman attending chama

Exclusion Criteria:

-

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Facility delivery | 22 months
  Proportion of women giving birth in a health facility based on questionnaire

SECONDARY OUTCOMES:
4 ANC visits | 22 months
  attendance at 4 or more ANC visits in pregnancy based on questionnaire
CHV homevisit | 22 months
  CHW homevisit within 48 hours of birth based on questionnaire
Exclusive breastfeeding | 22 months
  Initiation of solids to the infant after 6 months based on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Christoffersen-Deb, MDCM, Principal Investigator — Moi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maldonado LY, Songok JJ, Snelgrove JW, Ochieng CB, Chelagat S, Ikemeri JE, Okwanyi MA, Cole DC, Ruhl LJ, Christoffersen-Deb A. Promoting positive maternal, newborn, and child health behaviors through a group-based health education and microfinance program: a prospective matched cohort study in western Kenya. BMC Pregnancy Childbirth. 2020 May 12;20(1):288. doi: 10.1186/s12884-020-02978-w. PMID 32398156